CLINICAL TRIAL: NCT05733520
Title: I-CARE 2 RCT: Mobile Telehealth to Reduce Alzheimer'S-related Symptoms for Caregivers and Patients
Brief Title: I-CARE 2: Mobile Telehealth to Reduce Alzheimer'S-related Symptoms
Acronym: I-CARE 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Regenstrief Institute, Inc. (Other)
Responsible Party: Principal Investigator, Richard Holden, Department Chair, Dean's Eminent Scholar & Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15749; R01AG078234 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Caregiver Burden; Alzheimer Disease
Keywords: Alzheimer's disease and related dementias; Caregiver; Caregiver Burden; Behavioral and psychological symptoms of dementia
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease; Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the Brain CareNotes app or an attention control app.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary investigator and outcome assessor will be masked to the App assignment (Brain CareNotes vs Attention Control App)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain CareNotes App (Experimental)
  Interventions: Behavioral: Brain CareNotes
- Attention Control App (Active Comparator)
  Interventions: Behavioral: Dementia Guide Expert

INTERVENTIONS:
Behavioral: Brain CareNotes — The Brain CareNotes mobile telehealth app is used by unpaid caregivers for BPSD management. It includes remote communication with an external human support person-a care coach-as well as features for users to independently perform health-related activities.
  Arms: Brain CareNotes App
Behavioral: Dementia Guide Expert — Dementia Guide Expert provides education only and no interactive BPSD management support, coaching, assessment, or external response. It contains "evidence-based expert information on what dementia is, types, contributing factors, risks, symptoms, stages, diagnosis, tests, treatment, management, communication techniques, and links to resources and support services."
  Arms: Attention Control App

SUMMARY:
This study is a randomized, controlled trial (RCT) to evaluate the effect of Brain CareNotes (a mobile health application) on the burden experienced by unpaid caregivers of patients with dementia and on the behavioral and psychological symptoms of dementia (BPSD) displayed by care recipients. Over 39 months, the trial will enroll 184 caregivers of community-dwelling patients diagnosed with Alzheimer's disease or a related dementia (ADRD). Caregivers will be randomized to use the Brain CareNotes app or an attention control education-only app for 12 months, with usage reminders.

DETAILED DESCRIPTION:
This study is a hybrid efficacy-effectiveness RCT to evaluate the effect of Brain CareNotes on unpaid caregiver burden and patient BPSD. Over 39 months, the trial will enroll 184 caregivers. Participants will be randomized to use the Brain CareNotes app or an attention control education-only app (Dementia Guide Expert) for 12 months.

The primary objective is to test the effect of Brain CareNotes on a) caregiver burden and b) patient BPSD at 12 months. The investigators hypothesize that caregiver burden and patient BPSD will be lower among those participants randomized to the Brain CareNotes intervention compared to those randomized to the education-only attention control app at 12 months. The primary, powered outcomes are calculated using the caregiver-reported Neuropsychiatric Inventory (NPI); the total NPI score measures patient BSPD and the caregiver distress sub-score measures caregiver burden. The investigators will obtain NPI responses from caregivers at baseline, six, and 12 months.

The secondary objective is to test the effect of Brain CareNotes on a) caregiver depressive symptoms and b) patient and caregiver acute care utilization at 12 months. The investigators hypothesize that participants randomized to the Brain CareNotes intervention will have lower caregiver depressive symptoms and decreased acute care utilization compared to those randomized to the control app. For caregiver depressive symptoms, investigators will use the researcher-administered Patient Health Questionnaire-9 (PHQ-9) at baseline, six, and 12 months. Acute care utilization data will be obtained from self-reports or Indiana's statewide Health Information Exchange (HIE), known as the Indiana Network for Patient Care (INPC), to identify both caregivers' and patients' hospital and ER visits that occurred within 12 months of enrollment.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* Self-identified primary unpaid caregiver of a person diagnosed with ADRD (at any stage) who are:
* Receiving primary care and
* Community-dwelling;
* English literate;
* Age ≥ 18 years

Caregiver Exclusion Criteria:

* Care recipient is a permanent resident of an extended care facility (nursing home);
* Involvement in another clinical trial that would prevent or interfere with study objectives;
* Sensory or other impairment prohibiting the use of a mobile touchscreen device or other study activity (after correction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden | 12 months
  The burden experienced by caregivers caused by their caregiving responsibilities measured by the Neuropsychiatric Inventory (NPI) caregiver distress sub-score. The distress score is calculated by adding the distress score for each of the 12 items of the NPI. A score of 0 would indicate that the BPSD cause no distress while a score of 60 would indicate that each symptom causes severe distress for the caregiver.
Patient BPSD | 12 months
  Behavioral (e.g. agitation, aggression, wandering) and psychological (e.g. delusions, hallucinations) symptoms of dementia as measured by the Neuropsychiatric Inventory (NPI). The NPI is a 12-item questionnaire. The total score is calculated by adding the product of the frequency and severity of those 12 items. A score of 0 would indicate that no symptoms are present while a score of 144 would indicate that all symptoms are present at the highest level of frequency and severity.

SECONDARY OUTCOMES:
Caregiver Depressive Symptoms | 12 months
  Caregiver depression as measured by the Patient Health Questionnaire (PHQ)-9. The PHQ-9 is a 9-item questionnaire using a 0-3 rating scale. Scores range from 0-27. A total score of 0 represents no depression, while score of 5, 10, 15, and 20 serve as cut points for mild, moderate, moderately severe, and severe depression, respectively.
Caregiver Acute Care Utilization | 12 months
  Caregiver visits to emergency rooms, hospitals, or inpatient diagnoses. Obtained from caregiver self-reports or medical records.
Patient Acute Care Utilization | 12 months
  Patient visits to emergency rooms, hospitals, or inpatient diagnoses. Obtained from caregiver self-reports or medical records.

OTHER OUTCOMES:
Caregiver Self-efficacy | 12 months
  Caregiver perceived self-efficacy as measured using the Revised Scale for Caregiving Self-Efficacy. It consists of 3 sections each with five items. Participants rank self-efficacy on a scale of 0-100 for each item, with a higher score representing greater confidence. Thus, a high total score represents greater self-efficacy.
Caregiver Social Support | 12 months
  Caregiver perceived social support measured using the Multidimensional Scale of Perceived Social Support (MSPSS). The MSPSS is a 12-item questionnaire using a 7-point Likert scale where 1=very strongly disagree and 7=very strongly agree. Scores range from 12-84. A low score represents minimal social support while a high score represents a great level of perceived social support.
System Usability Scale | 12 months
  10-item standardized survey of user-reported technology usability, based on revised System Usability Scale, with scale score computed ranging from 0-100, with 100 indicating highest possible perceived usability.
Behavioral Intention Questionnaire | 12 months
  A 4-item questionnaire assessing a user's intention to use a technology in the near future. Scores range from 0-24 with a high score representing greater intention to use the technology.
App Use | 12 months
  Usage logs of app use over time.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Holden, PhD, Principal Investigator — Indiana University; Malaz Boustani, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - IU Health, Indianapolis, Indiana
  - Community Health Network, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No